CLINICAL TRIAL: NCT05957432
Title: Efficacy and Safety of Black Seed Oil With Vonoprazan Based Triple Therapy in Treatment of Helicobacter Pylori
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Alaa, clinical pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Black seed oil with Vonoprazan
Record Dates: First submitted 2023-06-16; First posted 2023-07-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; vonoprazan; black seed oil; oxidative stress
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 , Black seed oil group (Active Comparator): 45 patients will receive they will receive 1800 mg (4 soft gelatin capsules of 450 mg) black seed oil (2 capsules twice daily 30 min after the meal) for 6 weeks plus vonoprazan-based triple therapy ( conventional therapy ) consists of vonoprazan 20 mg twice daily, clarithromycin 500 mg twice daily, and amoxicillin 1000 mg twice daily for 14 days
  Interventions: Drug: Black Seed Oil Cap/Tab; Drug: Vonoprazan, Amoxicillin and Clarithromycin
- Group 2 , control group (Active Comparator): This group consists of 45 patients, who will receive vonoprazan-based triple therapy(conventional therapy ) consists of vonoprazan 20 mg twice daily, clarithromycin 500 mg twice daily, and amoxicillin 1000 mg twice daily for 14 days
  Interventions: Drug: Vonoprazan, Amoxicillin and Clarithromycin

INTERVENTIONS:
Drug: Black Seed Oil Cap/Tab — possessed anti-H. pylori activity comparable to triple therapy and improved dyspepsia symptoms in infected patients
  Other Names: Baraka 450 mg
  Arms: Group 1 , Black seed oil group
Drug: Vonoprazan, Amoxicillin and Clarithromycin — H pylori vonoprazan based treatment

SUMMARY:
The aim of this study is to:

• Evaluation of efficacy and safety of adding black seed oil with vonoprazan triple therapy ( vonoprazan ,clarithromycin and amoxicillin ) in eradication of Helicobacter pylori infection and this will be done through evaluation of:

A. Efficacy by:

1. determination of successful eradication,which will be considered to be achieved on the basis of a negative stool antigen test four weeks after the end of treatment using Stool Ag test
2. The effect of N. Sativa on:

I. Oxidative stress by measuring MDA II. Inflammation by measuring IL1B as inflammatory markers

B. Safety will be done through:

Monitoring of expected treatment related adverse effects (black seed oil and vonoprazan triple therapy ) will be done through the whole study period.

C. Symptoms evaluation using the Gastrointestinal symptom rating scale D. Assessment of patient's quality of life using SF36 questionnaire

DETAILED DESCRIPTION:
Helicobacter pylori infection is a highly prevalent chronic bacterial infection in humans worldwide affecting approximately 50% of the global population. H. pylori infection is highly prevalent in the Middle East and North Africa (MENA) region .

It may cause chronic gastritis, peptic ulcer disease, atrophic gastritis, and intestinal metaplasia that predispose to gastric cancer . Moreover, H. pylori may contribute to insulin resistance and metabolic syndrome as well as autoimmune and hematologic diseases . H. pylori was classified as a class I human carcinogen .

About 25 years ago, a proton pump inhibitor (PPI)-based regimen was introduced as a first-line treatment of H. pylori infection. PPI-based therapy showed a superior efficacy to non-PPI-based therapy in terms of H. pylori eradication.The PPI-based triple therapy, which consists of PPI, amoxicillin, and clarithromycin, has been a worldwide choice for H. pylori eradication. However, the treatment regimen is still a concern in light of the decreasing eradication rates owing to the increased antibiotic resistance of H. pylori.

Recently, vonoprazan, a novel potassium-competitive acid blocker, has been used in H. pylori eradication therapy in order to increase the eradication rate .

Vonoprazan (VPZ) works by competing for potassium on the luminal side of the parietal cell and causes rapid and reversible inhibition of H-K ATPase and therefore inhibits extended acid secretion. In contrast to PPIs, Vonoprazan is a more potent inhibitor of acid secretion. It has a rapid onset of action, less anti-secretory variability, greater safety, and better tolerability .

A meta-analysis of 10 studies by Jung et al. included research comparing the efficacy of a vonaprazan-based triple therapy group (vonoprazan 20 mg bid., amoxicillin 750 mg bid., and clarithromycin 200 or 400 mg bid. for 7 days) with that of a PPI-based triple therapy group (omeprazole 20 mg or lansoprazole 30 mg bid., amoxicillin 750 mg bid., and clarithromycin 200 or 400 mg bid. for 7 days). The eradication rates of vonoprazan-based triple therapy and PPI-based triple therapy were 87.9% and 72.8% (pooled risk ratio [RR] 1.02, 95% confidence interval [CI] 1.15-1.24), respectively.

The increasing rate of anti-H.Pylori drug resistance, medication costs, side effects, and the patient's incompliance make the treatment of H. pylori infection a global challenge. Therefore, there is a need to look for new safe, feasible, and affordable alternatives that are effective against H. pylori.

In recent years, the use of medicinal plants has been considered due to their potential effects on human health and the better management of diseases. Meanwhile, Nigella sativa is one of the most useful medicinal plants, which has been traditionally used for the treatment of many acute and chronic diseases and the promotion of human health.

The seeds of N. sativa, commonly known as black seed or black cumin, have rich biological active compounds such as thymoquinone (TQ), dithymoquinone, nigellicine, nigellidine, thymol, and carvacrol. All these compounds are synergistically responsible for beneficial pharmacological properties ; including antioxidant, anti-inflammatory, anticancer, antimicrobial, antiparasite, immunopotentiating action, gastroprotective, hepatoprotective, hypoglycemic, analgesic effects, and so forth.

In various studies, the antibacterial effects of this plant and its ingredients have been proven. The essential oil of N. sativa and its components like TQ and hydrothymoquinone were reported to be lethal to some Gram-negative and Gram-positive bacteria.

In an in vitro experiment, N. sativa extract inhibited the growth of all H. pylori strains within 60 min. The essential oil obtained from N. sativa was found to be safer than the volatile oil against different cell lines. Human case reports indicated allergic contact dermatitis following the use of some preparations containing N. sativa. However, clinical trials did not report any severe adverse effects following consumption N. sativa.

In a clinical trial, it was shown that N. sativa seed powder possessed anti-H. pylori activity comparable to triple therapy and improved dyspepsia symptoms in infected patients. It seems that the combination of N. sativa with antibiotics can reduce the resistance of H. pylori colonies and improve antibiotic efficacy.

H. pylori infection induces an inflammatory response that is also oxidative. The gastric epithelium and the bacteria induce production of interleukin-8 (IL-8) and malondialdehyde (MDA) that contributes to the generation of great amounts of toxic reactive oxygen species (ROS), with marked infiltration of inflammatory cells, and can elicit induction of interleukin-1β (IL-1β), interleukin-6 (IL-6), IL-8, interleukin-12 (IL-12), tumour necrosis factor-α (TNF-α) and interferon-γ (IFN-γ) .

IL-1β has biological effects that qualify it as arguably the most important cytokine in the gastrointestinal tract. Its proinflammatory properties contribute to the defence against pathogens, its antisecretory and cytoprotective effects contribute to the healing process following challenge to the integrity of the mucosa, and its acid inhibitory effects may have a profound effect on the natural history of H pylori infection.

Several studies have shown that NS has been proven to have antioxidant capabilities by reducing the production of reactive oxygen species (ROS), superoxide dismutase (SOD) and malondialdehyde (MDA).

Previous researches showed that supplementation of NS would significantly decrease the production of MDA and SOD in patients compared to controls.Interestingly, N. sativa Interestingly, TQ was found to exert its anti-inflammatory properties through the prevention of the expression of IL-6, IL-1β, and cyclooxygenase-2 in experimental rats.

No clinical trial has yet evaluated the effects of N. sativa oil concurrent with vonoprazan based regimens on the eradication of H. pylori infection. Therefore, The investigators performed this trial to evaluate the anti-H. Pylori properties of N. sativa concurrent with vonoprazan triple therapy on the eradication of bacteria, dyspepsia symptoms and quality of life in patients with this infection. Furthermore, the investigators measured the effects of N. sativa on oxidative stress and inflammatory markers in infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age 18 to 75 years old
* Patients with confirmed H. pylori infection by stool Ag test who had not received prior eradication therapy

Exclusion Criteria:

* History of hypersensitivity / allergy to any of the study drugs i.e., Esomeprazole, vonoprazan, penicillin, or clarithromycin
* History of previous H. pylori eradication therapy
* History of using PPIs, antibiotics that affect H. pylori within 4 weeks
* History of gastric malignancy or surgery
* Serious cardiovascular, pulmonary, renal, hepatic disorders or active malignancy
* Pregnancy or breast feeding
* History of drug abuse or active alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Stool antigen test at baseline ( pre-intervention) | at baseline for diagnosis of helicobacter pylori (before start of triple therapy )
  Stool Antigen Test: The test is qualitative and is based on the detection of H. pylori antigen in human feces ( positive test )
Change of Stool antigen test after 4 weeks from triple therapy | after 4 weeks from triple therapy
  evaluate successful eradication of helicobacter pylori by negative stool Ag test

SECONDARY OUTCOMES:
Change in MDA (oxidative stress marker) levels | change from baseline at 6 weeks
  For evaluating the effect of N. Sativa on oxidative stress analysis for measuring levels of MDA and IL_1B using ELISA Kits.
Change in Interleukin 1B ( inflammatory markers ) levels | change from baseline at 6 weeks
  effect of Nsativa on inflamatory markers
"Gastrointestinal symptom rating scale" | change from baseline at 6 weeks
  • Symptoms will be assessed using "Gastrointestinal symptom rating scale"GSRS is a validated GI questionnaire that utilises a 7-level Likert scale (1-7), based on the intensity and frequency of GI symptoms experienced during the previous seven days. A higher score represents the main symptoms complained about by the patients.
SF36 questionnaire | change from baseline at 6 weeks
  Quality of life of patients will be assessed using the SF36 questionnaire
Safety and tolerability | every week for 4 weeks
  Personal interviews with open-ended questions via questionnaire and self-reporting will be conducted by telephone every other day after enrollment in order to access adverse events and side effect
  The adverse effect that will be included in the questionnaire will be nausea, vomiting, bitter taste, skin rash, bloating, dizziness, headache, diarrhea, constipation, abdominal pain, and dry mouth or throat

CONTACTS AND LOCATIONS:
Overall Officials: sara M zaky, ass.prof, Principal Investigator — faculty of pharmacy Ain shams university; yasser A Elnaggar, prof, Study Chair — faculty of medicine zagazig university; sara F Mohamed, lecturer, Study Chair — faculty of pharmacy Ainshams university
Locations (1):
- GIT department zagazig university hospital, Zagazig, Egypt

REFERENCES:
- [Result] Sjomina O, Pavlova J, Niv Y, Leja M. Epidemiology of Helicobacter pylori infection. Helicobacter. 2018 Sep;23 Suppl 1:e12514. doi: 10.1111/hel.12514. PMID 30203587
- [Result] Wagner S, Varrentrapp M, Haruma K, Lange P, Muller MJ, Schorn T, Soudah B, Bar W, Gebel M. The role of omeprazole (40 mg) in the treatment of gastric Helicobacter pylori infection. Z Gastroenterol. 1991 Nov;29(11):595-8. PMID 1771934
- [Result] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775
- [Result] Suzuki S, Gotoda T, Kusano C, Iwatsuka K, Moriyama M. The Efficacy and Tolerability of a Triple Therapy Containing a Potassium-Competitive Acid Blocker Compared With a 7-Day PPI-Based Low-Dose Clarithromycin Triple Therapy. Am J Gastroenterol. 2016 Jul;111(7):949-56. doi: 10.1038/ajg.2016.182. Epub 2016 May 17. PMID 27185079
- [Result] Jung YS, Kim EH, Park CH. Systematic review with meta-analysis: the efficacy of vonoprazan-based triple therapy on Helicobacter pylori eradication. Aliment Pharmacol Ther. 2017 Jul;46(2):106-114. doi: 10.1111/apt.14130. Epub 2017 May 12. PMID 28497487
- [Result] Hashem-Dabaghian F, Agah S, Taghavi-Shirazi M, Ghobadi A. Combination of Nigella sativa and Honey in Eradication of Gastric Helicobacter pylori Infection. Iran Red Crescent Med J. 2016 Jun 21;18(11):e23771. doi: 10.5812/ircmj.23771. eCollection 2016 Nov. PMID 28191328
- [Result] Salem EM, Yar T, Bamosa AO, Al-Quorain A, Yasawy MI, Alsulaiman RM, Randhawa MA. Comparative study of Nigella Sativa and triple therapy in eradication of Helicobacter Pylori in patients with non-ulcer dyspepsia. Saudi J Gastroenterol. 2010 Jul-Sep;16(3):207-14. doi: 10.4103/1319-3767.65201. PMID 20616418
- [Result] Augusto AC, Miguel F, Mendonca S, Pedrazzoli J Jr, Gurgueira SA. Oxidative stress expression status associated to Helicobacter pylori virulence in gastric diseases. Clin Biochem. 2007 Jun;40(9-10):615-22. doi: 10.1016/j.clinbiochem.2007.03.014. Epub 2007 Mar 28. PMID 17466292
- [Result] Alizadeh-Naini M, Yousefnejad H, Hejazi N. The beneficial health effects of Nigella sativa on Helicobacter pylori eradication, dyspepsia symptoms, and quality of life in infected patients: A pilot study. Phytother Res. 2020 Jun;34(6):1367-1376. doi: 10.1002/ptr.6610. Epub 2020 Jan 9. PMID 31916648
- [Result] Kato M, Ota H, Okuda M, Kikuchi S, Satoh K, Shimoyama T, Suzuki H, Handa O, Furuta T, Mabe K, Murakami K, Sugiyama T, Uemura N, Takahashi S. Guidelines for the management of Helicobacter pylori infection in Japan: 2016 Revised Edition. Helicobacter. 2019 Aug;24(4):e12597. doi: 10.1111/hel.12597. Epub 2019 May 20. PMID 31111585
- [Result] Kouitcheu Mabeku LB, Bello Epesse M, Fotsing S, Kamgang R, Tchidjo M. Stool Antigen Testing, a Reliable Noninvasive Method of Assessment of Helicobacter pylori Infection Among Patients with Gastro-duodenal Disorders in Cameroon. Dig Dis Sci. 2021 Feb;66(2):511-520. doi: 10.1007/s10620-020-06219-0. Epub 2020 Apr 30. PMID 32350723
- [Result] Veijola L, Myllyluoma E, Korpela R, Rautelin H. Stool antigen tests in the diagnosis of Helicobacter pylori infection before and after eradication therapy. World J Gastroenterol. 2005 Dec 14;11(46):7340-4. doi: 10.3748/wjg.v11.i46.7340. PMID 16437639